CLINICAL TRIAL: NCT01315197
Title: Application of Massage for Low Back Pain in Nursing Staff
Brief Title: Massage for Low Back Pain in Nursing Staff
Acronym: Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Talita Pavarini Borges, University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Talita Pavarini Borges; Universidade de São Paulo (Other: Universidade de São Paulo)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2010-10

CONDITIONS: Low Back Pain
Keywords: Low back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Massage; Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- massage (Experimental): The massage Anma has Japanese origin and a protocol was used with smoothing, kneading and pressure points on the bladder meridian.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Massage Anmá: 7-8 sessions, twice per week, kneading and pressure points on the bladder meridian
  Other Names: Anmá; Oriental Massage; Acupressure

SUMMARY:
Objectives: Semi experimental Clinical Trial aimed at verifying the effectiveness of massage for lower back pain occupational as well as to assess the influence of technique in performing work activities and life in the team nursing.

DETAILED DESCRIPTION:
Method: 18 officials received 7-8 massage sessions, twice per week, with the same protocol points. Data were collected on baseline, after one and two months and they responded 2 questionnaires (Functional Assessment of Oswestry and Risk Assessment in Movement and Transfer Scale) and the Numeric Pain Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the study of employees with availability of time for submission to the sessions
2. Not be pregnant
3. Hold shift of at least 6 hours daily
4. Do not go on vacation or leave care during the study period
5. Reporting back pain self-reported or confirmed by medical diagnosis
6. Not having passed off due to back pain in past 6 months
7. Do not submit spondylolisthesis, disc herniation and sciatic pain self-reported or confirmed by medical diagnosis
8. Do not use anti-inflammatory drugs
9. Individuals that showed greater than 0 (zero) in the Numerical Pain Scale (10) Score higher than 15 on the Functional Assessment Questionnaire Oswestry

Exclusion Criteria:

* Employees who left the study or that lost more than one session

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Application of Massage for Low Back Pain in Nursing Staff | two months
  Effectiveness of massage in alleviating lower back pain through response to 2 questionnaires (Functional Assessment of Oswestry and Risk Assessment in Movement and Transfer Scale) and the Numeric Pain Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Talita P Borges, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Borges TP, Greve JM, Monteiro AP, da Silva RE, Giovani AM, da Silva MJ. Massage application for occupational low back pain in nursing staff. Rev Lat Am Enfermagem. 2012 May-Jun;20(3):511-9. doi: 10.1590/s0104-11692012000300012. English, Portuguese, Spanish. PMID 22991113